CLINICAL TRIAL: NCT03509207
Title: A Pilot Study of Peroral Vorinostat (SAHA) in Patients With Refractory Histone Deacetylase-positive Uterine Sarcoma
Brief Title: Vorinostat (SAHA) in Uterine Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The early termination was NOT due to safety reasons, terminated because of the very slow recruitment and problematic access to the study medication in Europe
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHA
Record Dates: First submitted 2018-03-27; First posted 2018-04-26 (Actual); Results first posted 2020-07-27 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Leiomyosarcoma; Endometrial Stromal Tumors; Carcinosarcomas Uterine
Keywords: Uterine sarcoma; Histone deacetylases
MeSH Terms: conditions — Leiomyosarcoma; Endometrial Stromal Tumors | interventions — Vorinostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vorinostat, Zolinza Oral Capsules (Experimental): Vorinostat Oral Capsules 400mg daily
  Interventions: Drug: Vorinostat Oral Capsule

INTERVENTIONS:
Drug: Vorinostat Oral Capsule — Vorinostat, 400 mg orally once daily for the first 14 days of a 21 day cycle Treatment will be continued for 4 cycles. Patients with a response or stable disease after 4 cycles will be continued on vorinostat therapy at the tolerated schedule and dosage until disease progression, unacceptable toxicity or patients' withdrawal of the consent. At the maximum, a total of 12 cycles will be administered over a period of 9 months.
  Other Names: Zolinza

SUMMARY:
Uterine sarcomas are rare tumors with a poor prognosis.

The main purpose of this phase II proof-of-principle- pilot study is to test the efficacy of the hydroxamic acid-based Histone deacetylase inhibitor (HDACI) Vorinostat (SAHA) as monotherapy in patients with HDAC-positive, progressive, metastatic uterine sarcomas and mixed epithelial and mesenchymal tumors after prior anti-proliferative therapy.

DETAILED DESCRIPTION:
This is an open-label, single arm, proof of concept-study of the HDAC-inhibitor vorinostat in patients with refractory uterine sarcoma that have been pre-tested for an high expression of HDAC. Patients will receive Vorinostat, 400 mg (4 capsules á 100mg of Zolinza) orally once daily for the first 14 days of a 21 day cycle. Treatment will be continued for 4 cycles (treatment period 1). Patients with a response or stable disease after 4 cycles as determined by computed tomography (CT) of target an non target-lesions will be continued on vorinostat therapy at the tolerated schedule and dosage until disease progression, unacceptable toxicity or patients' withdrawal of the consent. At the maximum, a total of 12 cycles will be administered over a 9 months period (treatment periods 2 and 3).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic uterine sarcoma (endometrial stromal sarcoma, undifferentiated uterine sarcoma, leiomyosarcoma, adenosarcoma and carcinosarcoma

  * High HDAC-positivity of the tumor determined by immunohistochemistry
  * Patients must have received prior systemic antineoplastic therapy
  * Patient is not amenable for curative therapy
  * Age >= 18 years
  * Estimated life expectancy > 3 months
  * Measurable disease on CT/MRI (at least one measurable lesion >1cm) or chest X-ray (at least one measurable lesion >2cm)
  * Karnofsky performance status of 60-100
  * Adequate hematologic, renal and hepatic function
  * Subject is able to swallow and retain oral medication and does not have uncontrolled emesis
  * No fertility preserved
  * Written informed consent

Exclusion Criteria:

* Lack of or low expression of HDAC (see 4.1 "Pre-Screening")

  * Significant cardiac disease
  * Other invasive malignant tumor diagnosed within the last 5 years (e.g. metastases from breast cancer in the last 3 years)
  * Significant bowel obstruction
  * Severe uncontrolled infection
  * Known HIV-positivity
  * Symptomatic brain metastasis or leptomeningeal disease
  * Pre-existing significant liver disease, severe hepatic impairment (Bilirubin no greater than 1.5 times upper limit of normal (ULN) and/or aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) greater than 2.5 times ULN)
  * Known history of allergic reaction to vorinostat or similar medications
  * Systemic therapy or an investigational agent within 21 days prior to study inclusion
  * Uncontrolled hypertension (sustained systolic blood pressure > 150 mmHg or diastolic pressure > 100 mmHg despite optimal medical management)
  * Major surgery within 3 weeks of enrollment when diagnosed at an early stage
  * Symptomatic congestive heart failure
  * Unstable angina pectoris or cardiac arrhythmia
  * Myocardial infarction within last 6 months
  * Known active hepatitis B or hepatitis C
  * Psychiatric illness/social situations that would limit compliance with study requirements-
  * Prior history of thrombotic or thromboembolic events, unless adequately controlled by anticoagulant therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigated condition occurs exclusively in women
Enrollment: 3 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Petru, MD, Principal Investigator — Department of OB/GYN of the Medical University of Graz
Locations (1):
- Medical University of Graz, Clinic of Obstetrics and Gynecology, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 patients were enrolled. The study was prematurely closed due to the sluggish patient recruitment and the difficult acquisition of the investigational product.
Pre-assignment Details: There were no Screening failures in the Course of the study.
Period: Overall Study
Arm/Group | Vorinostat, Zolinza Oral Capsules
Started | 3
Completed | 1
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Statistical evaluation was not possible as only 1 Patient reached end point 1.
Arm/Group | Vorinostat, Zolinza Oral Capsules
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Change from Baseline Tumor Size to last available observation with respect to progress as defined by RECIST 1.1 (CT-Scan every 12 weeks up to 9 months)
Time Frame: 9 months
Population: Only one Patient reached the first end Point. Statistical Evaluation was therefore not possible. For this reason no data are reported in the data table.
Arm/Group | Vorinostat, Zolinza Oral Capsules
Number analyzed (Participants) | 0

2. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: This endpoint is evaluated by the amount of clinical adverse experiences.
Time Frame: 9 months
Population: as for outcome 1
Arm/Group | Vorinostat, Zolinza Oral Capsules
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From enrolment to study completion per Patient, up to 41 weeks.
Arm/Group | Vorinostat, Zolinza Oral Capsules
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat, Zolinza Oral Capsules (N=3)
Death of uterine carcinoma (Reproductive system and breast disorders) | 2 (2)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
abscess of the vaginal vault (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT03509207/Prot_000.pdf